CLINICAL TRIAL: NCT02258230
Title: Laparoscopic 3D Versus 2D Sacral Colpopexy and Paravaginal Repair for Pelvic Organ Prolapse: a Comparison of Operative Times and Complications
Brief Title: Laparoscopic Three-dimensional Versus Two-dimensional Sacral Colpopexy and Paravaginal Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Collaborators: International Urogynecology Associates (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4859
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Pelvic Organ Prolapse; Cystocele
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2D mode LSC (Active Comparator): 2D mode of the 3D Laparoscopic Video System for the Laprascopic Sacral Colpopexy (LSC) arm. Use of the 3D laparoscopic system can be switched to either 2D or 3D.
  Interventions: Device: 2D mode of the 3D Laparoscopic Video System
- 3D mode LSC (Active Comparator): 3D mode of the 3D Laparoscopic Video System for the Laprascopic Sacral Colpopexy (LSC) arm. Use of the 3D laparoscopic system can be switched to either 2D or 3D.
  Interventions: Device: 3D mode of the 3D Laparoscopic Video System
- 2D mode PVR (Active Comparator): 2D mode of the 3D Laparoscopic Video System for the Paravaginal Repair (PVR) arm. Use of the 3D laparoscopic system can be switched to either 2D or 3D.
  Interventions: Device: 2D mode of the 3D Laparoscopic Video System
- 3D mode PVR (Active Comparator): 3D mode of the 3D Laparoscopic Video System for the Paravaginal Repair (PVR) arm. Use of the 3D laparoscopic system can be switched to either 2D or 3D.
  Interventions: Device: 3D mode of the 3D Laparoscopic Video System

INTERVENTIONS:
Device: 3D mode of the 3D Laparoscopic Video System — Olympus 3DV-190 3D Visualization Unit. LTF-190-10-3D: ENDOEYE FLEX 3D Videoscope.
  Arms: 3D mode LSC; 3D mode PVR
Device: 2D mode of the 3D Laparoscopic Video System — Olympus 3DV-190 3D Visualization Unit. LTF-190-10-3D: ENDOEYE FLEX 3D Videoscope.
  Arms: 2D mode LSC; 2D mode PVR

SUMMARY:
Compare operative times and complications of sacral colpopexy and paravaginal repair between two-dimensional and three-dimensional laparoscopic systems.

DETAILED DESCRIPTION:
The purpose of this study is to compare operative times of laparoscopic sacral colpopexy (LSC) for the treatment of symptomatic vaginal vault prolapse as well as paravaginal repair (PVR) for symptomatic cystocele between two-dimensional and three-dimensional laparoscopic systems. Additionally this study will evaluate postoperative complications from surgeries performed using two-dimensional versus three-dimensional laparoscopic systems.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic vaginal vault prolapse (stage 2 or greater point C-1 pelvic organ prolapse quantification [POP-Q] or grade 2 or greater Baden-Walker half way system) undergoing laparoscopic sacral colpopexy

And/Or

* Symptomatic cystocele (stage 2 or greater, point Aa or Ba > -1 POP-Q or grade 2 or greater Baden-Walker half way system) undergoing laparoscopic paravaginal repair

Exclusion Criteria:

* Age less than 18 years
* Inability to comprehend questionnaires
* Inability to give informed consent or to return for review
* Vaginal vault prolapse < stage 2
* Unable to undergo general anesthesia
* More than 5 previous laparotomies
* Prior sacral colpopexy or vaginal mesh prolapse procedure
* Prior surgery involving the retropubic space
* Vaginal length less than 6 cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Operative Times | Intraoperative
  Operative times of laparoscopic sacral colpopexy and paravaginal repair procedures from the first part of dissection until closure of the peritoneum.

SECONDARY OUTCOMES:
Complications | Intraoperative up to 6 weeks post procedure
  Intraoperative complications will be recorded. Post operative complications will be reported for the first 6 weeks after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Moore, DO, Principal Investigator — International Urogynecology Associates
Locations (2):
- United States (2):
  - Beverly Hills Sunset Surgery Center, Los Angeles, California
  - Northside Hospital, Atlanta, Georgia

REFERENCES:
- See also: International Urogynecology Associates' website — http://www.miklosandmoore.com/